CLINICAL TRIAL: NCT06726421
Title: Systemic Therapy Combined With Radiotherapy Versus Systemic Therapy Alone for Oligometastatic Kidney CancER (STROKER): A Multicenter, Randomized Controlled Phase III Trial
Brief Title: Systemic Therapy Alone or With Stereotactic Body Radiotherapy for Oligometastatic Kidney Cancer (STROKER Study)
Acronym: STROKER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-FXY-190; B2024-536-01 (Other: Sun Yat-sen University Cancer Center Clinical Research Center)
Record Dates: First submitted 2024-11-22; First posted 2024-12-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer); Kidney Cancer Metastatic; Renal Cell Carcinoma Metastatic
Keywords: radiotherapy; SBRT; SABR; oligometastatic; oligometastasis
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Radiosurgery; Sunitinib; pazopanib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT arm (Experimental): Patients undergo SBRT to all metastatic sites in addition to standard systemic therapy. Patients should complete radiotherapy for all lesions within 6 months of enrollment, preferably within the first 3 months.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT); Drug: axitinib ± immune checkpoint inhibitors (ICIs), lenvatinib ± ICIs, cabozantinib ± ICIs, sunitinib and pazopanib
- Control arm (Active Comparator): Patients receive standard systemic therapy.
  Interventions: Drug: axitinib ± immune checkpoint inhibitors (ICIs), lenvatinib ± ICIs, cabozantinib ± ICIs, sunitinib and pazopanib

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — The preferred treatment plan is SBRT with a fraction dose ≥7 Gy. The prescription dose should ensure a BED of no less than 115. Radiotherapy is usually delivered daily, every other day, or other interval decided by treating radiation oncologist.
  Other Names: Stereotactic ablative radiotherapy
  Arms: SBRT arm
Drug: axitinib ± immune checkpoint inhibitors (ICIs), lenvatinib ± ICIs, cabozantinib ± ICIs, sunitinib and pazopanib — Standard systemic therapy are targeted agents or their combination with immunotherapy recommended by guidelines. This may include axitinib ± immune checkpoint inhibitors (ICIs), lenvatinib ± ICIs, cabozantinib ± ICIs, sunitinib and pazopanib, etc.
  Other Names: Standard systemic therapy

SUMMARY:
This phase III randomized controlled trial evaluates the efficacy of stereotactic body radiation therapy (SBRT) in oligometastatic renal cell carcinoma. The study aims to determine if the addition of SBRT to standard systemic therapy prolong survival compared to the standard systemic therapy alone. In addition, the study will explore the impact of this combined modality therapy on patients' toxicity and quality of life. The researchers will compare SBRT plus standard systemic therapy to standard systemic therapy alone, which is targeted agents and immunotherapy in this case, to determine if SBRT could prolong survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To compare the progression-free survival (PFS) between patients receiving SBRT + standard systemic therapy versus standard systemic therapy alone.

SECONDARY OBJECTIVES:

I. To compare the overall survival (OS) between patients receiving SBRT + standard systemic therapy versus standard systemic therapy alone.

II. To compare the cancer specific survival (CSS) between patients receiving SBRT + standard systemic therapy versus standard systemic therapy alone.

III. To estimate the local control (LC) rate of SBRT. IV. To compare the post-treatment progression-free survival (post-treatment PFS) between patients receiving SBRT + standard systemic therapy versus standard systemic therapy alone.

V. To evaluate treatment-related toxicity after adding SBRT based on patient-reported outcomes and researcher reported adverse events.

VI. To compare the quality of life between patients treated with SBRT or not using EQ-5D-5L, FKSI-DRS and FKSI-19.

OUTLINE: Patients are randomized to either Control arm or SBRT arm.

Control arm: Patients receive standard of care systemic therapy on study. SBRT arm: Patients undergo SBRT to all metastatic sites in addition to standard of care systemic therapy on study.

Patients periodically receive computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI) throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of renal cell carcinoma of any histology
* Age ≥ 18 years.
* ECOG performance status of 0-2.
* Imaging suggests the presence of distant metastases, with no more than 5 metastatic lesions according to RECIST 1.1 criteria and MDA standards.
* The patient has received local therapy to primary site, including surgery, stereotactic radiotherapy, or ablation.
* The patient has received no more than 2 lines of systemic therapy.
* No significant impairment of major organ function:

Hemoglobin (HB) ≥ 80 g/L Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L Platelets (PLT) ≥ 75 × 10⁹/L Serum total bilirubin ≤ 1.5 × ULN Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN

Exclusion Criteria:

* Presence of intracranial metastases.
* Target lesions have previously received high-dose irradiation with .
* Target lesions are unsuitable for radiation therapy judged by treating radiation oncologist (e.g., lesions invading the gastrointestinal tract or penetrating the bronchus).
* Uncontrollable metastatic pleural effusion or ascites.
* Presence of other malignancies that have not been cured.
* History of significant psychiatric disorders that impede understanding of informed consent and compliance with the study protocol.
* Presence of other serious illnesses that may pose significant risks or affect radiation therapy.
* Women who are pregnant, breastfeeding, or with plans for childbearing during the study.
* Any other reasons deemed by the investigator to make the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From enrollment to disease progression, up to 5 years
  the time from randomization to the first occurrence of tumor progression or death. If no progression occurs, PFS is measured up to the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival | From enrollment to death from any cause, up to 5 years
  The time from randomization to death from any cause. If no death occurs, OS is measured up to the date of the last follow-up.
Cancer specific survival | From enrollment to death from cancer, up to 5 years
  the interval from randomization to death caused by renal cancer. If no death occurs, it is measured up to the date of the last follow-up.
Local control rate | From enrollment to in-field progression, up to 5 years
  The interval from randomization to progression of each SBRT treatment lesion. If no progression occurs, it is measured up to the date of the last follow-up.
Post-treatment progression free survival | From the initiation of systemic treatment to disease progression, up to 5 years
  The time from the initiation of systemic treatment for metastasis to the first occurrence of tumor progression or death after enrollment. If no progression occurs, it is measured up to the date of the last follow-up.
Progression-free survival 2 | From the initiation of systemic treatment to disease progression, up to 5 years
  Defined as the time from randomization to progression on the next-line treatment or death from any cause.
Incidence of Adverse Events | Up to 2 years
  Adverse events need to be grouped and analyzed based on treatment-related events, including all grades and grades 3-4 events. Adverse events are assessed by investigators according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Patient-Reported Adverse Events | Up to 2 years
  Adverse events will be selected from the patient-reported outcomes (PRO) scoring system developed by the National Cancer Institute (NCI) for toxic events (specifically, the NCI PRO-CTCAE™ ITEMS Chinese version). These items will be provided to patients, who will self-assess and report any adverse events experienced during each treatment cycle.
Health-related quality of life by EQ-5D-5L | Up to 2 years
  The overall quality of life will be evaluated using the European Quality of Life 5-Dimension 5-Level (EQ-5D-5L) scale.
Health-related quality of life by FSKI | Up to 2 years
  For assessing quality of life related to advanced kidney cancer, the Functional Assessment of Cancer Therapy - Kidney Cancer Symptom Index (FKSI), developed by the American Outcomes Research and Education Center, will be utilized, which includes both the FKSI-DRS and FKSI-19 scales.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Union Hospital, Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No